CLINICAL TRIAL: NCT03869814
Title: Non-invasive Liquid Biopsy Analysis of Epigenomics Signatures in Multiple Cancer Types
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ClearNote Health (Industry)
Responsible Party: Sponsor
Other Study IDs: MT1410
Record Dates: First submitted 2019-03-05; First posted 2019-03-11 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Diagnosis of Cancer of Various Organs
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Non-cancer: 3,250 asymptomatic individuals without prior history of cancer
  Interventions: Other: Blood Draw
- Cancer: 3,250 individuals with confirmed malignancy
  Interventions: Other: Blood Draw

INTERVENTIONS:
Other: Blood Draw — Blood Draw

SUMMARY:
Bluestar Genomics is developing a test from whole blood for the early detection of multiple cancers. The goal of this study is to employ genomics, epigenomics and proteomics methodology for the detection of cancer signal in the blood of subjects with solid tumors. The study will include subjects without cancers that will be followed up every 6-months for up to 3-years from blood draw.

DETAILED DESCRIPTION:
Epigenomic changes in cancer cells can provide a rich source of biomarker signals for the detection of disease. As cancer cells manifest their epigenomic changes in blood due to cell death, DNA and protein molecules can be probed using specific molecular analytic approaches. Bluestar Genomics employs epigenomic technologies to measure dynamic changes in DNA demethylation events via direct measurement of 5-hydroxymethyl-cytosine residues in cfDNA. Companion assays are also run to provide information on cfDNA digestion patterns and protein-based changes in plasma. This information, combined in a machine learning framework, enable the provision of prediction models that report on the presence of cancer and the determination of the tissue of tumor origin. This study will build predictive models and test performance of these models to detect the presence of cancer and tissue of origin in several cancer type by using a matched case-control study design.

ELIGIBILITY:
Inclusion Criteria

1. Subjects must be between 45 - 75 years of age at the time of enrollment
2. Patient fully consented
3. Cancer diagnosis OR high clinical suspicion for cancer, based on the participating site's and practitioner's standards of care (SOC)
4. No previous history of cancer and treatment naïve at time of enrollment

Exclusion Criteria

1. Age < 45 OR > 75 years of age
2. Any prior cancer diagnosis with or without treatment (with the exception of non-melanoma skin cancers resolved/treated > 1 year prior to enrollment)
3. Receipt of any cancer therapy including chemotherapy, radiation, palliative radiation, hormonal or naturopathic therapies
4. In situ carcinoma without an invasive component
5. Any surgery requiring general anesthesia within 2 months of collection. Anesthesia used in procedures such as colonoscopy and EBUS is acceptable.
6. Dental Novocain within 1 week of collection
7. Receipt of systemic immunomodulation therapy within past 12 months
8. Currently pregnant, or pregnancy within last 12 months
9. Organ transplantation
10. Received dialysis
11. Blood transfusion within 1 month
12. HIV/AIDs, Hepatitis A, D, or E, TB, any kind of prion disorder (e.g., CJD) or other infectious pathogens currently present or present in past 5 years.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Both study groups enrolled at medical centers across the United States
Sampling Method: Non-Probability Sample
Enrollment: 6500 (Estimated)
Dates: Start 2018-04-05 (Actual); Primary Completion 2023-06-13 (Estimated); Study Completion 2023-09-13 (Estimated)

PRIMARY OUTCOMES:
Detection of cancer signal in the cancer cohort | 1 year
  Evaluation of genomics, proteomic and epigenomics signals, such as 5-hydroxymethylcytosine (5hmC), contained in plasma, in comparison to these signals in plasma from non-cancer controls
Detection of tissue of origin signal in the cancer cohort | 1 year
  Evaluation of genomics, proteomic and epigenomics signals, such as 5-hydroxymethylcytosine (5hmC), contained in plasma, in comparison to these signals from non-cancer controls

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Levy, Ph.D., Study Director — ClearNote Health
Locations (1):
- Bluestar Genomics, Inc., San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No